CLINICAL TRIAL: NCT05116228
Title: Randomized, Prospective, Active-comparator Controlled, Patient-blinded Study to Demonstrate Non-inferiority of Reduced-dose Rituximab in Rheumatoid Arthritis Patients in Low Disease Activity and Remission - the REDOREM Study
Brief Title: Non-inferiority of Reduced-dose Rituximab in Rheumatoid Arthritis in Low Disease Activity and Remission
Acronym: REDOREM
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Failure to recruit
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Peter Mandl, Co-Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-002156-27
Record Dates: First submitted 2018-03-21; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Rheumatoid Arthritis; Remission
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 500mg RTX Group (Active Comparator): Patients in this group will receive 1x500mg (500mg RTX group) RTX (Mabthera) at baseline (time-point of their upcoming semi-annual infusion) and at months 6, 12, 18 and 24
  Interventions: Drug: 500mg RTX Group
- 1000mg RTX group (Active Comparator): Patients in this group will receive 1x1000mg RTX (Mabthera) at baseline (time-point of their upcoming semi-annual infusion) and at months 6, 12, 18 and 24
  Interventions: Drug: 1000mg RTX Group

INTERVENTIONS:
Drug: 500mg RTX Group — Patients will receive 1x500mg RTX (Mabthera) at baseline (time-point of their upcoming semi-annual infusion) and at months 6, 12, 18 and 24
  Other Names: Mabthera 500mg
  Arms: 500mg RTX Group
Drug: 1000mg RTX Group — Patients will receive 1x1000mg RTX (Mabthera) at baseline (time-point of their upcoming semi-annual infusion) and at months 6, 12, 18 and 24
  Other Names: Mabthera 1000mg
  Arms: 1000mg RTX group

SUMMARY:
To investigate whether a reduced-dose dosing regimen (1x500mg semiannually) of rituximab (RTX) (Mabthera®) is non-inferior in patients with rheumatoid arthritis (RA) whose disease is in persistent low disease activity (LDA) or clinical remission (REM) (pLDA/pREM) as compared to the standard dosing regimen of 1x1000mg semi-annual infusions.

DETAILED DESCRIPTION:
Randomized, controlled, single-centre study with 1x500mg or 1x1000 semi-annual infusions of RTX (Mabthera) as intervention and a follow-up period of 2 years. Patients as well as assessors will be blinded to the type of treatment. Patients in the 1x500mg group who experience a flare as defined by the disease activity score 28-ESR (DAS28) will receive 1x1000mg RTX (Mabthera) at their upcoming scheduled infusion appointment. Patients in the 1x1000mg group whose disease activity reaches DAS28 >3.2 during the duration of the study will be re-evaluated for a change in biological therapy and will discontinue the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA according to the 2010 American College of Rheumatology (ACR) / European League Against Rheumatism (EULAR) classification criteria
* Current treatment with RTX (at time of inclusion have already received at least 2 cycles of 1000mg RTX) at the Day-Clinic of the Division of Rheumatology of the Medical University of Vienna
* Persistent low disease activity or clinical remission as defined below
* Persistent clinical remission (pREM) will be defined as a simplified disease activity index (CDAI) (12) ≤2.8 measured at two time-points 6 months apart. The CDAI is calculated as follows: tender joint count (TJC) + swollen joint count (SJC) + patient's assessment of general health on a 100 mm visual analogue scale (GH) + evaluator's assessment of general health on a 100 mm visual analogue scale (EGH)
* Persistent low disease activity (pLDA) will be defined as a CDAI ≤10 measured at two timepoints 6 months apart Patients who achieve REM at only either one of the two successive time-points will be considered as having pLDA with regard to the current trial

Exclusion Criteria:

* Patients ≤ 18 yrs
* Patients receiving RTX for a disease other than RA
* Patients who fail to meet criteria for REM or LDA at either one of the two successive timepoints (i.e. having a disease activity >10 as measured by the clinical disease activity index, (CDAI))

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-09-01; Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Proportion of flare | month 24
  Disease activity score 28-Erythrocyte sedimentation sate (DAS28-ESR), Scale 0 (best) - 10 (worse)

SECONDARY OUTCOMES:
Radiographic progression | month 12
  Sharp modified van der Heijde (SvdH) score, Scale 0 (best) - 488 (worse)
Radiographic progression | month 24
  Sharp modified van der Heijde (SvdH) score, Scale 0 (best) - 488 (worse)
Physical function | months 12
  Health assessment questionnaire disability index (HAQ-DI), Scale 0 (best) - 3.0 worse
Physical function | months 24
  Health assessment questionnaire disability index (HAQ-DI), Scale 0 (best) - 3.0 worse
Proportion of flare | month 21
  Disease activity score 28-Erythrocyte sedimentation sate (DAS28-ESR), Scale 0 (best) - 10 (worse)
Proportion of flare | month 18
  Disease activity score 28-Erythrocyte sedimentation sate (DAS28-ESR), Scale 0 (best) - 10 (worse)
Proportion of flare | month 15
  Disease activity score 28-Erythrocyte sedimentation sate (DAS28-ESR), Scale 0 (best) - 10 (worse)
Proportion of flare | month 12
  Disease activity score 28-Erythrocyte sedimentation sate (DAS28-ESR), Scale 0 (best) - 10 (worse)
Proportion of flare | month 9
  Disease activity score 28-Erythrocyte sedimentation sate (DAS28-ESR), Scale 0 (best) - 10 (worse)
Proportion of flare | month 6
  Disease activity score 28-Erythrocyte sedimentation sate (DAS28-ESR), Scale 0 (best) - 10 (worse)
Proportion of flare | month 3
  Disease activity score 28-Erythrocyte sedimentation sate (DAS28-ESR), Scale 0 (best) - 10 (worse)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No